CLINICAL TRIAL: NCT03849495
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of CKD-370 With D745 in Healthy Volunteers
Brief Title: Pharmacokinetics and Safety/Tolerability After Oral Administration of CKD-370 and D745 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 191BE18033
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): * Period 1: D745
  * Period 2: CKD-370
  Interventions: Drug: CKD-370; Drug: D745
- Group B (Experimental): * Period 1: CKD-370
  * Period 2: D745
  Interventions: Drug: CKD-370; Drug: D745

INTERVENTIONS:
Drug: CKD-370 — Test drug
Drug: D745 — Reference drug

SUMMARY:
A randomized, open-label, single dose, two-way crossover study to compare the pharmacokinetics and safety/tolerability of CKD-370 with D745 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years
2. Females who are not pregnant or breastfeeding or who have surgical infertility
3. Signed informed consent form
4. Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

1. History of clinically significant hepatic, renal, nervous, immune, respiratory, digestive, urinary, endocrine, hemato-oncology, cardiovascular systemic disease or psychosis disorder
2. Clinical laboratory test values are outside the accepted normal range at Screening

   * aspartate aminotransferase(AST), alanine aminotransferase(ALT) > 1.5 times the upper limit of the normal range
   * Total Bilirubin > 1.5 times the upper limit of the normal range
   * creatine phosphokinase(CPK) > 1.5 times the upper limit of the normal range
   * estimated Glomerular Filtration Rate(eGFR, MDRD* formula) < 60 mL/min/1.73m2 (*MDRD: Modification of Diet in Renal Disease)
   * Positive reaction on following tests: Hepatitis B, Hepatitis C, human immunodeficiency virus(HIV) and syphilis
   * systolic blood pressure(SBP) ≥ 150 mmHg or < 90 mmHg, diastolic blood pressure(DBP) > 100 mmHg or < 50 mmHg
3. Current smokers or those who cannot quit smoking during the period from 90 days before the first IP dosing to the last discharge.
4. Subject who drink excessive caffeine or alcohol continuously and who cannot discontinue caffeine or alcohol intake during the period from 3 days before the first IP dosing to the last discharge.
5. Participated in a clinical trial within 90 days prior to first IP dosing
6. Not eligible to participate for the study at the discretion of Investigator
7. Other exclusive inclusion criteria, as defined in the protocol

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-03-17 (Estimated); Study Completion 2019-03-21 (Estimated)

PRIMARY OUTCOMES:
AUClast of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Empagliflozin
Cmax of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Maximum plasma concentration of Empagliflozin

SECONDARY OUTCOMES:
AUCinf of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Empagliflozin
Tmax of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Time to maximum plasma concentration of Empagliflozin
T1/2 of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Half-life of Empagliflozin
CL/F of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Apparent clearance of Empagliflozin
Vd/F of Empagliflozin | 0 hour ~ 48 hour after drug administration
  Apparent volume of distribution of Empagliflozin

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, Ph.D. M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea